CLINICAL TRIAL: NCT02208544
Title: Efficacy of [18F]-2-fluoro-2-deoxy-D-glucose Positron Emission Tomography (FDG-PET) in Evaluation of Cytological Indeterminate Thyroid Nodules Prior to Surgery: a Multicentre Cost-effectiveness Study
Brief Title: FDG-PET/CT in Evaluation of Cytological Indeterminate Thyroid Nodules to Prevent Unnecessary Surgery (EfFECTS)
Acronym: EfFECTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: KUN 2014-6514; NL50166.091.14 (Registry Identifier: ToetsingOnline)
Record Dates: First submitted 2014-07-22; First posted 2014-08-05 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-02

CONDITIONS: Thyroid Nodule; Thyroid Neoplasms
Keywords: Thyroid Nodule; Indeterminate Cytology; FDG-PET/CT; Diagnostic Thyroid Surgery; Efficacy; Cost-Effectiveness; Quality-of-Life; Thyroidectomy
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms | interventions — Thyroidectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FDG-PET/CT-driven (Experimental): Following treatment based on FDG-PET/CT:
  * negative: watchful waiting including confirmatory ultrasound
  * positive: diagnostic thyroid surgery as planned
  Interventions: Procedure: Diagnostic Thyroid Surgery; Device: Ultrasound of the head and neck; Radiation: FDG-PET/CT
- Current Practice (Other): diagnostic thyroid surgery despite results of FDG-PET/CT
  Interventions: Procedure: Diagnostic Thyroid Surgery; Radiation: FDG-PET/CT

INTERVENTIONS:
Procedure: Diagnostic Thyroid Surgery — Diagnostic Thyroid Surgery
  Other Names: Thyroid Lobectomy; Hemithyroidectomy; Thyroidectomy
Device: Ultrasound of the head and neck — Confirmatory Neck Ultrasonography in FDG-PET/CT negative patient in the experimental arm
  Arms: FDG-PET/CT-driven
Radiation: FDG-PET/CT — Head and Neck FDG-PET/CT
  Other Names: fluorodeoxyglucose positron emission tomography

SUMMARY:
The purpose of this study is to determine whether the use of molecular imaging using FDG-PET/CT could prevent unnecessary diagnostic thyroid surgery in case of indeterminate cytology during fine-needle aspiration biopsy.

DETAILED DESCRIPTION:
Rationale: Only about ¼ of patients with thyroid nodules with indeterminate cytology are proven to suffer from a malignancy at diagnostic hemithyroidectomy. Therefore ~¾ is operated upon unbeneficially. Recent studies using FDG-PET/CT have suggested that it can decrease the fraction of unbeneficial procedures from ~73% to ~40%. Thereby the direct costs per patient, the number of hospitalization and average sick leave days might decrease and the experienced HRQoL might increase. A study will be undertaken to show the additional value of FDG-PET/CT after indeterminate cytology with respect to unbeneficial procedures, costs and utilities.

Main objective: To determine the impact of FDG-PET/CT on decreasing the fraction of patients with cytologically indeterminate thyroid nodules undergoing unbeneficial patient management.

Study design: A prospective, multicentre, randomized, stratified controlled blinded trial with an experimental study-arm (FDG-PET/CT-driven) and a control study-arm (diagnostic hemithyroidectomy, independent of FDG-PET/CT-result).

Study population: Adult patients with a cytologically indeterminate thyroid nodule, without exclusion criteria, in 15 (university and regional) hospitals distributed over the Netherlands.

Intervention: One single FDG-PET/low-dose non-contrast enhanced CT of the head and neck is performed in all patients. Patient management depends on allocation and results of this FDG-PET/CT.

Main study parameters/endpoints: The number of unbeneficial interventions, i.e. surgery for benign disease or watchful-waiting for malignancy.

Secondary objectives: complication rate, consequences of incidental PET-findings, number of hospitalisation and sick leave days, volumes of healthcare consumed, experienced health-related quality-of-life (HRQoL), genetic, cytological and (immuno)histopathological features of the nodules.

Sample size calculation/data analysis: Based on above-mentioned estimated reduction in unbeneficial interventions from ~73% to ~40%, at least 90 patients with nodules>10 mm need to be analyzed (2:1 allocation, α=0.05, power=0.90, single-sided Fisher's exact test). After correction for nodule size and data-attrition, 132 patients need to be included in total. Intention-to-treat analysis will be performed. Incremental Net Monetary Benefit based on the total direct costs per patients and the gain in HRQoL-adjusted survival years are computed. Cytological, histological and genetic parameters for FDG-avidity will be described.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All patients undergo one FDG-PET/CT scan of head/neck (effective dose: <3.5 mSv) and are asked to fill in 6 questionnaires at 4 timepoints. FDG-PET/CT negative patients in the experimental arm will undergo a single confirmatory US (±FNAC). An interim/posterior analysis of the control subjects is performed to ensure oncological safety. In case of an unexpected high false-negative ratio in this control arm, all patients will be advised to undergo surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Documented history of a solitary thyroid nodule or a dominant nodule within multinodular disease, with (US-guided) FNAC performed by a dedicated radiologist or experienced endocrinologist or pathologist, demonstrating an indeterminate cytological examination (i.e. Bethesda category III or IV) according to the local pathologist and confirmed after central review;
2. Scheduled for surgical excision (preferably) within 2 months of the inclusion date;
3. Age ≥ 18 years;
4. Euthyroid state with a serum thyrotropin (TSH) or a free T4 level within the institutional upper and lower limits of normal, measured within 2 months of registration. In case of a suppressed TSH: a negative 123I, 131I or 99mTcO4- scintigraphy must be available ("cold nodule");
5. In patients with multinodular disease and a dominant nodule, the nuclear medicine physician responsible for FDG-PET/CT scan interpretation must determine whether the nodule is likely to be discriminated on FDG-PET/CT imaging prior to enrolment;
6. Willing to participate in all aspects of the study;

Exclusion Criteria:

1. High a priori probability of malignancy:

   * FNAC Bethesda category V or VI during local reading or central review;
   * Prior radiation exposure / radiotherapy to the thyroid;
   * Prior neck surgery or radiation that in the opinion of the PI has disrupted tissue architecture of the thyroid;
   * New unexplained hoarseness, change of voice, stridor or paralysis of a vocal cord;

     * In case a benign reason has been found (e.g. vocal cord edema), the patient is eligible;
   * Thyroid nodule discovered as a FDG-PET positive incidentaloma
   * New cervical lymphadenopathy highly suspicious for malignancy;

     * In case malignancy is excluded, patient is eligible;
   * Previous treatment for thyroid carcinoma or current diagnosis of any other malignancy that is known to metastasize to the thyroid;
   * Known metastases of thyroid carcinoma;
   * Known genetic predisposition for thyroid carcinoma:

     * Familiar Non-Medullary Thyroid Cancer (NMTC)
     * Familiar Papillary Thyroid Cancer (FPTC)
     * Familiar Adenomatoid Polyposis Coli syndrome (FAP, Gardner syndrome, APC-gene mutations on chromosome 5q21)
     * Morbus Cowden (PTEN mutation on chromosome 10q23.3)
     * PTC / nodular thyroid hyperplasia / papillary renal tumours. Linked to locus 1q21.
2. Proven benign disease or insufficient material for a cytological diagnosis:

   * FNAC Bethesda category I or II during local reading or central review
3. Performance of non-routine additional diagnostic tests that alter the patients treatment policy (e.g. mutation analysis on cytology)
4. Inability to undergo randomization:

   * Any patient that will receive thyroid surgery for other reasons (e.g. mechanical or cosmetic complaints).
5. Inability to undergo treatment:

   * Inability to undergo surgery in the opinion of the surgeon / anaesthetist.
6. Contra-indications for FDG-PET/CT:

   * Patient has evidence of infection localized to the neck in the 14 days prior to the FDG-PET/CT scan;
   * Inability to tolerate lying supine for the duration of an FDG-PET/CT examination (~10-15min);
   * Poorly regulated diabetes mellitus (see next item);
   * Hyperglycaemia at time of FDG injection prior to PET/CT (fasting serum glucose >200mg/dL [>11.1 mmol/L]);

     * The use of short-acting insulins within 4 hours of the PET scan is not allowed
   * If female and fertile: signs and symptoms of pregnancy or a positive pregnancy test / breast-feeding;

     * A formal negative pregnancy test is not obligatory
   * (severe) claustrophobia;

     * Low dose benzodiazepines are allowed
7. General contra-indications:

   * Inability to give informed consent;
   * Severe psychiatric disorder;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Fraction of unbeneficial treatment | 12 months after inclusion
  Unbeneficial treatment is defined as either:
  * surgery in benign disease
  * watchful waiting in malignant disease
  benign or malignant disease is defined on final histology (after surgery) or 12 month follow-up including confirmatory neck ultrasonography.
  This parameter is compared between both study arms based on intention-to-treat.

SECONDARY OUTCOMES:
Fraction Complications | 12 months after inclusion
  SO1b: To determine the effect of incorporation of FDG-PET/CT on the complication-ratio.
Fraction False-Negative FDG-PET/CT's | 12 months after inclusion
  SO1c: To determine the false-negative fraction of FDG-PET/CT in this population.
Lesion and Patient Characteristics | 12 months after inclusion
  SO1d: To determine the influence of lesion size, pathological classification and patient characteristics on the diagnostic accuracy of FDG-PET/CT.
Fraction Incidental FDG-PET/CT Findings | 12 months after inclusion
  SO1e: To determine whether incorporation of FDG-PET/CT of the head and neck lead to overdiagnosis in non-thyroidal incidental findings.
Overall and Disease Free Survival | 12 months after inclusion
  SO1f: To determine the short-term overall and disease free survival in both study arms.
FDG-PET/CT Implementation-hampering Factors | 12 months after inclusion
  SO1g: To determine which factors hamper implementation of this modality for this indication (structured interviews).
Fraction of Patients being operated despite negative FDG-PET/CT | 12 months after inclusion
  SO1h: To determine the fraction of patients that cannot be reassured by a negative PET-scan (experimental arm only) despite careful selection of patients (implementability).
HRQoL-scores according to SF36-II, EQ-5D-5L, SF-HLQ and ThyPRO including changes | Baseline, 2 months, 6 months and 12 months after inclusion
  SO2a: To determine the impact on the experienced HRQoL between the group with and without FDG-PET/CT according to 4 different questionnaires at 4 timepoints during the first 12 months after FDG-PET/CT.
  SO2b: To determine whether patients in the experimental arm with negative PET-findings have a different HRQoL than those who receive surgery independent of the FDG-PET/CT results.
Direct Costs | 12 months after inclusion
  SO3a: To determine the effect of incorporation of FDG-PET/CT on the mean direct costs (=volume of care multiplied by activity based costs) per patient during the first 12 months after FDG-PET/CT.
Number of Hospitalisation Days | 12 months after inclusion
  SO3b: To determine the effect of incorporation of FDG-PET/CT on the average length of hospital stay for treatment of (complications of) thyroid lesions?
Number of Sick Leave Days | 3 months after inclusions
  SO3c: To determine the total number of sick leave days for the first three months in the patients? Do these differ between both study arms?
incremental Net Monetary Benefit | 12 months after inclusion
  SO3d: To determine the incremental Net Monetary Benefit of incorporation of FDG-PET/CT with respect to quality-adjusted life-years (QALYs, based on EQ-5D-5L index and overall survival) saved including sensitivity analysis.
  SO3e: To determine the incremental Net Monetary Benefit of incorporation of FDG-PET/CT with respect to decrease in unbeneficial treatment.
  Sensitivity analysis will be performed. A mere description will be given as there is no "accepted" value for this kind of analysis.
Tissue Protein- and Gene-expression profile | 12 months after inclusion of last patient
  SO4a: Are there potential protein- or gene-expression profiles, capable of determining the nature of the FNAC-indeterminate nodes (cytology) SO4b: What is the interaction/correlation between the parameters mentioned in SO4a and the results of the FDG-PET/CT scan and the final diagnosis?
Molecular biomarkers in relation to FDG-PET/CT | 12 months after inclusion of last patient
  SO4b: What is the interaction/correlation between the parameters mentioned in SO4a and the results of the FDG-PET/CT scan and the final diagnosis?
  * Can these tissue molecular biomarkers help in selecting the patients that benefit most from FDG-PET, or vice versa?
  * Can higher pre-operative diagnostic accuracy be achieved by combining FDG-PET and molecular biomarkers?
  * Are molecular biomarkers related to false-positive or false-negative FDG-PET/CT results?

CONTACTS AND LOCATIONS:
Overall Officials: Lioe-Fee de Geus-Oei, MD, PhD, Study Chair — Leiden University Medical Center, Leiden, the Netherlands; Dennis Vriens, MD, PhD, Study Director — Leiden University Medical Center, Leiden, the Netherlands; Lisanne de Koster, MD, Principal Investigator — Radboud University Medical Centre, Nijmegen, the Netherlands
Locations (15):
- Netherlands (15):
  - Radboudumc, Nijmegen, Gelderland
  - MUMC, Maastricht, Limburg
  - AMC, Amsterdam, North Holland
  - VUmc, Amsterdam, North Holland
  - LUMC, Leiden, South Holland
  - ErasmusMC, Rotterdam, South Holland
  - MeanderMC, Amersfoort, Utrecht
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Rijnstate, Arnhem
  - Reinier de Graaf Ziekenhuis, Delft
  - UMCG, Groningen
  - St. Antonius, Nieuwegein
  - HagaZiekenhuis, The Hague
  - UMCU, Utrecht
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and datasets generated during and/or analysed during the current study are available from the corresponding author on reasonable request. Data requestors will need to sign a data access agreement and in keeping with patient consent for secondary use, obtain ethical approval for any new analyses.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting 2023.
Access Criteria: The study protocol and datasets generated during and/or analysed during the current study are available from the corresponding author on reasonable request. Data requestors will need to sign a data access agreement and in keeping with patient consent for secondary use, obtain ethical approval for any new analyses.

REFERENCES:
- [Background] de Geus-Oei LF, Pieters GF, Bonenkamp JJ, Mudde AH, Bleeker-Rovers CP, Corstens FH, Oyen WJ. 18F-FDG PET reduces unnecessary hemithyroidectomies for thyroid nodules with inconclusive cytologic results. J Nucl Med. 2006 May;47(5):770-5. PMID 16644746
- [Background] Vriens D, de Wilt JH, van der Wilt GJ, Netea-Maier RT, Oyen WJ, de Geus-Oei LF. The role of [18F]-2-fluoro-2-deoxy-d-glucose-positron emission tomography in thyroid nodules with indeterminate fine-needle aspiration biopsy: systematic review and meta-analysis of the literature. Cancer. 2011 Oct 15;117(20):4582-94. doi: 10.1002/cncr.26085. Epub 2011 Mar 22. PMID 21432844
- [Background] Vriens D, Adang EM, Netea-Maier RT, Smit JW, de Wilt JH, Oyen WJ, de Geus-Oei LF. Cost-effectiveness of FDG-PET/CT for cytologically indeterminate thyroid nodules: a decision analytic approach. J Clin Endocrinol Metab. 2014 Sep;99(9):3263-74. doi: 10.1210/jc.2013-3483. Epub 2014 May 29. PMID 24873995
- [Background] de Koster EJ, de Geus-Oei LF, Dekkers OM, van Engen-van Grunsven I, Hamming J, Corssmit EPM, Morreau H, Schepers A, Smit J, Oyen WJG, Vriens D. Diagnostic Utility of Molecular and Imaging Biomarkers in Cytological Indeterminate Thyroid Nodules. Endocr Rev. 2018 Apr 1;39(2):154-191. doi: 10.1210/er.2017-00133. PMID 29300866
- [Result] de Koster EJ, de Geus-Oei LF, Brouwers AH, van Dam EWCM, Dijkhorst-Oei LT, van Engen-van Grunsven ACH, van den Hout WB, Klooker TK, Netea-Maier RT, Snel M, Oyen WJG, Vriens D; EfFECTS trial study group. [18F]FDG-PET/CT to prevent futile surgery in indeterminate thyroid nodules: a blinded, randomised controlled multicentre trial. Eur J Nucl Med Mol Imaging. 2022 May;49(6):1970-1984. doi: 10.1007/s00259-021-05627-2. Epub 2022 Jan 4. PMID 34981165
- [Result] de Koster EJ, Noortman WA, Mostert JM, Booij J, Brouwer CB, de Keizer B, de Klerk JMH, Oyen WJG, van Velden FHP, de Geus-Oei LF, Vriens D; EfFECTS trial study group. Quantitative classification and radiomics of [18F]FDG-PET/CT in indeterminate thyroid nodules. Eur J Nucl Med Mol Imaging. 2022 Jun;49(7):2174-2188. doi: 10.1007/s00259-022-05712-0. Epub 2022 Feb 9. PMID 35138444
- [Derived] de Koster EJ, Morreau H, Bleumink GS, van Engen-van Grunsven ACH, de Geus-Oei LF, Links TP, Wakelkamp IMMJ, Oyen WJG, Vriens D. Molecular Diagnostics and [18F]FDG-PET/CT in Indeterminate Thyroid Nodules: Complementing Techniques or Waste of Valuable Resources? Thyroid. 2024 Jan;34(1):41-53. doi: 10.1089/thy.2023.0337. Epub 2023 Dec 28. PMID 38009209
- [Derived] de Koster EJ, Vriens D, van Aken MO, Dijkhorst-Oei LT, Oyen WJG, Peeters RP, Schepers A, de Geus-Oei LF, van den Hout WB; EfFECTS trial study group. FDG-PET/CT in indeterminate thyroid nodules: cost-utility analysis alongside a randomised controlled trial. Eur J Nucl Med Mol Imaging. 2022 Aug;49(10):3452-3469. doi: 10.1007/s00259-022-05794-w. Epub 2022 Apr 18. PMID 35435497